CLINICAL TRIAL: NCT04027270
Title: Pelvic Health and Physical Therapy to Improve Lives of Prostate Cancer Patients
Brief Title: Pelvic Health and Physical Therapy to Improve Lives of Prostate Cancer Patients Undergoing Prostatectomy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jennifer Y Stone, Manager, Clinical Rehabilitative Services, University of Missouri-Columbia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015982
Record Dates: First submitted 2019-07-02; First posted 2019-07-19 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomization into treatment and standard of care groups. Treatment group will receive physical therapy in addition to standard of care treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): These individuals will receive standard of care for post operative recovery following a prostatectomy.
- Physical Therapy (Experimental): These individuals will receive post operative physical therapy in addition to standard of care for post operative recovery following a prostatectomy.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — Physical therapy 1-2 times per week for 3 months postoperatively to include lifestyle education, manual therapy, and exercise.
  Arms: Physical Therapy

SUMMARY:
Patients will be randomized into standard of care or receiving pre and post operative physical therapy intervention following prostatectomy. Outcome measures will be gathered to assess impact of physical therapy on function and quality of life.

DETAILED DESCRIPTION:
This is a prospective, randomized, non-blinded, research study undergoing robotic-assisted laparoscopic prostatectomy at the University of Missouri/Ellis Fischel Hospital. Participants will be randomized in a 1:1 fashion. Data also will be tracked on those who are post-operatively stratified by cancer grade and addition of radiation therapy (XRT) as XRT after surgery is dependent on participant pathology therefore would not be able to be determined in advance.

The study will be broken up into four phases, as described in detail below:

Phase 1:

* Urologic oncology team will consist of a urologic oncologist/surgeon, urologic nurse, and oncology nurse navigator practicing in a specialty oncology hospital which is part of a large regional hospital network in the Midwest section of the United States. A pelvic health physical therapist will be an additional member of this team practicing primarily in outpatient based clinics affiliated with a with the same large regional hospital network.
* Enrollment will be offered during first hospital visit with urologic oncology team confirming diagnosis of prostate cancer in and decision for robotic radical prostatectomy. Enrollment goal will be at least 40 men but caps at 100.
* The capture of participants for enrollment will be limited to a 12 month period.
* Consent is obtained and the participant is enrolled
* At the time of enrollment, all participants will have baseline measurements taken to obtain baseline physical assessment, complete baseline quality of life questionnaires, and receive education on exercises to begin as prehabilitation protocol prior to surgical intervention.

  o Baseline questionnaires include:
  1. International Prostate Symptom Score (IPSS)
  2. International Index of Erectile Function (IIEF)
  3. National Institute of Health Chronic Prostatitis Symptom Index (NIH-CPSI)
  4. Pain Visual Analog Scale (VAS)
  5. Beck's Depression Index (BDI)
  6. Bristol Stool Form Scale (BSFS)
* After obtaining written consent, subjects will be randomized to receive post-operative pelvic health physical therapy (Rehab group) or no post-operative intervention (control).
* Both groups will be given pre-operative prehabilitative exercise program and education of continence behavioral training.
* At the time of enrollment, all participants the will receive the same educational packet and home exercise program education from the urologic oncology team.

  o Home exercise (prehabilitative) protocol: transverse abdominus activation training, deep diaphragmatic breathing, urinary continence behavioral training and training for pelvic floor muscle proper activation using cues of "shorten the penis" for isolation of the muscles of urinary continence and "tighten around the anus" for posterior pelvic floor activation.
* Perioperative care, surgery and anesthesia, for all subjects will be per standard hospital protocol

Phase 2

* At the preoperative visit (1-2 week prior to surgery), both Rehab and Control group participants will meet with a physical therapist who specializes in orthopedic and pelvic health interventions.
* Control group will not meet with a physical therapist at the preoperative visit.

  o No additional education, teaching or rehabilitative intervention will be implemented outside of enrollment visit for the control group
* Objective measurements to be assessed by pelvic health physical therapist may include: Pelvic floor observation (ability to contract, relax and resting tone); pelvic floor manual muscle testing (MMT) for strength assessment using internal and RUSI measuring power, endurance and "quick flick ability"; abdominal wall mobility and scar/incision mobility (once adequately healed); core muscle activation mechanics and strength (including transverse abdominus, oblique and rectus abdominus); breathing mechanics; trigger point and tender point assessment of pelvic floor, pelvic girdle and abdominal wall; hip and lumbar spine screening for mobility, flexibility and posture; squat mechanics; balance of lower extremity; hip flexor, hamstring, psoas, gastrocnemius and solues tissue flexibility.
* Subjective measurements to be assessed by pelvic health physical therapist may include: pain rating, number of pads/diapers used daily, sexual activity and function, bowel consistency and frequency, urinary urgency and frequency, and level of urinary incontinence or leakage.
* Participant will see physical therapist 1 time total prior to surgery to review deficit areas, review pelvic floor muscle activation/strengthening exercises and educate on expected deficits post-prostatectomy.
* Radical robotic prostatectomy (RALP) will be performed by Urologic Oncologist. If the surgical intervention plan is altered so that participant is no longer eligible for RALP or additional surgical interventions are needed, participant will be excluded from further study enrollment and hence dismissed from study.
* Participant will be discharged from hospital based on surgeon discretion and appropriateness. Foley catheter will stay in place 14 days (+/- 7 days).

Phase 3

* Post-operative outpatient physical therapy program will begin within 1 week of Foley catheter removal after surgery for those randomly assigned to the Rehab group.
* Only the Rehab group participants will meet with a physical therapist who specializes in orthopedic and pelvic health interventions, Control group will do no formal physical therapy.
* Control group will be administered repeat baseline questionnaires via email, mail or phone call.
* Re-evaluation of all baseline measurements and questionnaires will be repeated for the randomly assigned Rehab group and implementation of customized exercise plans to improve post-operative deficit areas will begin.

  o Outpatient physical therapy intervention may include but not be limited to spinal stabilization activities, pelvic floor muscle re-education using digital/proprioceptive training as well as rehabilitative ultrasound imaging (RUSI), manual therapy (scar/myofascial mobilization), patient education and urinary continence behavioral training.
* Biofeedback training will be utilized with digital/manual and RUSI only; there will be no passive internal probe biofeedback based training utilized in this study.
* Rehab group participants will be seen by the same physical therapist once a week for 12 weeks (8-12 sessions, 45 minutes each).
* Appropriate re-evaluative objective and subjective measurements will be taken at 6 weeks post-operatively and 12 weeks post-operatively during final physical therapy visit.

Phase 4:

* During the 3 month follow-up with urologic oncology team, a pelvic health physical therapist will re-assess baseline subjective and objective measurements for Control groups and Rehab group as needed (if not obtained at 12 week final physical therapy visit).
* Both Rehab group and Control groups will be given repeat baseline questionnaires at 3 month follow-up.
* Participants will follow up with urologic oncologist and nurse navigator for regular prostate cancer check-ups at 2 weeks, 6 weeks, 12 weeks, 6 months, 9 months, 12 months, 18 months and 24 months post-operatively.
* During the 6 month, 9 month, 12 month 18 month and 24 month follow-ups with urologic oncology team, a pelvic health physical therapist will re-assess baseline subjective and objective measurements for both the Rehab and Control groups. Participants will re-complete baseline questionnaires at each visit.
* Both Rehab group and Control groups will be given repeat baseline questionnaires at the 6 month, 9 month, 12 month 18 month and 24 month follow-ups with urologic oncology team
* All research and demographic data will be collected and stored in secure EMR (electronic medical records) and REDCap (Research Electronic Data Capture) database
* Research data will be analyzed as appropriate by a medical research assistant using:

  * One-way analysis of variance (ANOVA)
  * T-tests
  * Fischer's exact
  * Wilcoxon Rank Sum Test
  * Generalized Estimation Equation (GEE) model

Criteria for participant eligibility:

Subject Population

- Undergoing RALP University of Missouri/Ellis Fischel Hospital for prostate cancer

Subject Inclusion

* Age greater than or equal to 18 years
* Men who have prostate cancer (regardless of grade or metastasis)
* Robotic assisted RALP performed by Urologic Oncologist
* Fluent in speaking and understanding English

Subject Exclusion

* Inability to obtain written informed consent
* Atrioventricular conduction blocks
* CV instability and concomitant use of alpha agonists or beta blockers
* Recent myocardial infarction (≤ 6 months ago)
* Cardiac arrhythmia disorders
* Stokes-Adams syndrome
* Wolff-Parkinson-White syndrome
* Seizure disorders
* Liver failure or hepatic dysfunction
* Significant renal disease with a serum creatinine ≥ 2 mg/dl
* A family history of malignant hyperthermia
* Current use of opioids or documented history of opioid abuse
* Unavailability for reliable transportation
* Typically, have less than 3 bowel movement per week
* Combined surgical cases that include robotic prostatectomy
* Non-fluent in English speaking and understanding

RECRUITMENT PLAN Participants will be recruited from the practices of the Division of Urologic Oncology, Department of Surgery at the University of Missouri/Ellis Fischel Hospital. The study will be introduced to every eligible patient scheduled for robot assisted laparoscopic prostatectomy by the participating consenting urologic oncologist from the Department of Surgery-Urology Division and a written consent obtained prior to surgery by the consenting research personnel. Candidate subjects will be provided time to consider the study, to read the informed consent document at their convenience, and discuss the study with family and others, as desired.

PRETREATMENT EVALUATION This study does not require any additional pretreatment evaluations other than those which are part of current clinical care standards for a patient undergoing RALP at University of Missouri. Preoperative evaluations follow recommendations from the NICE.47, 48

For RALP these include:

* Routine history and physical examination to include documentation of any comorbidities, medications (including complementary and alternative medications), family history, social history (alcohol and tobacco usage), height, body weight, Karnofsky performance status within 30 days of surgery
* Chest X-ray or CT scan of the Chest within 30 days of surgery
* Pre-operative laboratory investigations: CBC, BMP, urinalysis (dipstick, microalbumin, creatinine, microscopic evaluation if indicated), urine culture if indicated within 30 days of surgery
* Baseline EKG

SURGICAL INTERVENTION PLAN The technique of surgery will be robotic assisted laparoscopy based on the discretion of the surgeon and participant. None of the techniques utilized in the study are considered experimental and all are considered standard therapeutic options for the patient with prostate cancer concerning for cancer amenable to prostatectomy, respectively. Participant medications will be recorded from the home medications list and managed perioperatively per institutional standards.

The operating team will consist of the Medical Director and Urologic Oncologist on faculty at University of Missouri Department of Surgery-Urology Division. The procedures are performed under standardized general anesthesia with standard intraoperative vital sign monitoring.

EVALUATION DURING TREATMENT/INTERVENTION This protocol does not require any additional evaluations after the subject is admitted for surgery other than those routinely part of clinical care for a patient undergoing robot assisted laparoscopic prostatectomy other than inquiring for subjects' satisfaction on postop day one and monitoring for signs severe adverse effects during inpatient hospitalization. If severe adverse effects are suspected the appropriate treatment will be given per the standard of care at University of Missouri/Ellis Fischel Hospital.

Routine evaluation and management for those undergoing robot assisted laparoscopic prostatectomy include:

* ASA classification, assigned by the anesthesiologist
* Deep venous thrombosis prophylaxis per standardized pathway
* Estimated blood loss
* Use of intraoperative fluids (crystalloid, colloid, blood products)

CRITERIA FOR THERAPEUTIC RESPONSE/OUTCOME ASSESSMENT If the surgery is aborted for any reason before attempted excision of the mass fails for any reason, the participant will be removed from the study and replaced. Based on past experience these issues are rare events. If any robotic procedure converts to an open procedure, the participant will be excluded from the study. The postoperative period is defined as the period from the extubation to the study endpoint at 24 month post-operatively.

CRITERIA FOR REMOVAL FROM STUDY Participants will be withdrawn from the study if a desire is expressed to do so, if it is determined to be in the participant's best interest to do so, or if the individual does not undergo initiation of their surgical procedure as stipulated previously. If surgery is converted from robotic assisted to open the subject will be excluded from analysis. Occurrence of new cancer onset, or metastasis that requires additional surgical intervention or unpredicted treatments, participants will be withdrawn from the study. Participants who are not evaluable for the study primary endpoint by failure to obtain data for the primary endpoint will be excluded from the study and further analysis will not be performed.

ELIGIBILITY:
Inclusion Criteria:

* - Age greater than or equal to 18 years
* Men who have prostate cancer (regardless of grade or metastasis)
* Robotic assisted RALP performed by Urologic Oncologist
* Fluent in speaking and understanding English

Exclusion Criteria:

* - Inability to obtain written informed consent
* Atrioventricular conduction blocks
* CV instability and concomitant use of alpha agonists or beta blockers
* Recent myocardial infarction (≤ 6 months ago)
* Cardiac arrhythmia disorders
* Stokes-Adams syndrome
* Wolff-Parkinson-White syndrome
* Seizure disorders
* Liver failure or hepatic dysfunction
* Significant renal disease with a serum creatinine ≥ 2 mg/dl
* A family history of malignant hyperthermia
* Current abuse of opioids or documented history of opioid abuse
* Unavailability for reliable transportation
* Combined surgical cases that include robotic prostatectomy
* Non-fluent in English speaking and understanding

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
International Prostate Symptom Score Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in IPPS from preoperative through to 18 months post operatively, assessed at intervals
International Index of Erectile Function Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in IIEF from preoperative through to 18 months post operatively, assessed at intervals
National Institute of Health Chronic Prostatitis Symptom Index Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in NIH-CPSI from preoperative through to 18 months post operatively, assessed at intervals
Pain Visual Analog Scale Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in Pain VAS from preoperative through to 18 months post operatively, assessed at intervals
Beck's Depression Index Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in BDI from preoperative through to 18 months post operatively, assessed at intervals
Bristol Stool Scale Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in Bristol Stool Scale from preoperative through to 18 months post operatively, assessed at intervals
Pelvic Floor Strength Test Change | Preoperatively, 3 months post operatively, 9 months post operatively, 12 months post operatively, 18 months post operatively
  Change in strength from preoperative through to 18 months post operatively, assessed at intervals

CONTACTS AND LOCATIONS:
Locations (1):
- Jennifer Stone, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nam RK, Cheung P, Herschorn S, Saskin R, Su J, Klotz LH, Chang M, Kulkarni GS, Lee Y, Kodama RT, Narod SA. Incidence of complications other than urinary incontinence or erectile dysfunction after radical prostatectomy or radiotherapy for prostate cancer: a population-based cohort study. Lancet Oncol. 2014 Feb;15(2):223-31. doi: 10.1016/S1470-2045(13)70606-5. Epub 2014 Jan 17. PMID 24440474
- [Result] Wallis CJ, Herschorn S, Saskin R, Su J, Klotz LH, Chang M, Kulkarni GS, Lee Y, Kodama RT, Narod SA, Nam RK. Complications after radical prostatectomy or radiotherapy for prostate cancer: results of a population-based, propensity score-matched analysis. Urology. 2015 Mar;85(3):621-7. doi: 10.1016/j.urology.2014.11.037. PMID 25733275
- [Result] Pedraza R, Nieto J, Ibarra S, Haas EM. Pelvic muscle rehabilitation: a standardized protocol for pelvic floor dysfunction. Adv Urol. 2014;2014:487436. doi: 10.1155/2014/487436. Epub 2014 Jun 11. PMID 25006337
- [Result] Hung HC, Hsiao SM, Chih SY, Lin HH, Tsauo JY. An alternative intervention for urinary incontinence: retraining diaphragmatic, deep abdominal and pelvic floor muscle coordinated function. Man Ther. 2010 Jun;15(3):273-9. doi: 10.1016/j.math.2010.01.008. Epub 2010 Feb 24. PMID 20185357
- [Result] Ribeiro LH, Prota C, Gomes CM, de Bessa J Jr, Boldarine MP, Dall'Oglio MF, Bruschini H, Srougi M. Long-term effect of early postoperative pelvic floor biofeedback on continence in men undergoing radical prostatectomy: a prospective, randomized, controlled trial. J Urol. 2010 Sep;184(3):1034-9. doi: 10.1016/j.juro.2010.05.040. PMID 20643454